CLINICAL TRIAL: NCT05932615
Title: Evaluation of the Navitor Transcatheter Heart Valve in Low and Intermediate Risk Patients Who Have Severe, Symptomatic, Aortic Stenosis Requiring Aortic Valve Replacement
Brief Title: ENVISION IDE Trial: Safety and Effectiveness of NAVITOR in Transcatheter Aortic Valve Implantation
Acronym: ENVISION
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABT-CIP-10487
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-09

CONDITIONS: Aortic Valve Stenosis; Heart Valve Diseases; Aortic Valve Disease; Heart Disease Structural Disorder
Keywords: NAVITOR; Heart disease; Transcatheter aortic valve implantation (TAVI); Aortic stenosis; Cardiovascular diseases
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Valve Diseases; Aortic Valve Disease; Heart Diseases; Cardiovascular Diseases | interventions — Transcatheter Aortic Valve Replacement; Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Navitor Transcatheter Aortic Valve Implantation (TAVI) System (Experimental): TAVI with Abbott Navitor Transcatheter Aortic Valve Implantation (TAVI) System
  Interventions: Device: Navitor Transcatheter Aortic Valve Implantation (TAVI) System
- Any Commercially Available Transcatheter Aortic Valve System (CAV) (Active Comparator): TAVI with any FDA approved commercially available Transcatheter Aortic Valve System (CAV)
  Interventions: Device: Any Commercially Available Transcatheter Aortic Valve (CAV) System

INTERVENTIONS:
Device: Navitor Transcatheter Aortic Valve Implantation (TAVI) System — TAVI for relief of calcific aortic stenosis in patients with symptomatic heart disease who are at intermediate or low risk for open surgical therapy.
  Arms: Navitor Transcatheter Aortic Valve Implantation (TAVI) System
Device: Any Commercially Available Transcatheter Aortic Valve (CAV) System — TAVI for relief of calcific aortic stenosis in patients with symptomatic heart disease who are at intermediate or low risk for open surgical therapy.
  Arms: Any Commercially Available Transcatheter Aortic Valve System (CAV)

SUMMARY:
The objective of ENVISION is to evaluate the safety and effectiveness of the Navitor Transcatheter Aortic Valve Implantation (TAVI) System for treating patients with symptomatic, severe native aortic stenosis who are considered intermediate or low risk for surgical mortality.

The trial will also evaluate the safety and effectiveness of the Navitor TAVI System in a valve-in-valve (ViV) application in patients with symptomatic heart disease due to failure of a surgical or transcatheter bioprosthetic aortic valve who are at high or greater surgical risk.

DETAILED DESCRIPTION:
ENVISION is a prospective, multi-center clinical investigation at up to 115 sites globally. The objective of this clinical investigation is to evaluate the safety and effectiveness of the Navitor TAVI System for treating patients with symptomatic, severe native aortic stenosis who are considered intermediate or low risk for surgical mortality. The trial will register subjects in two separate cohorts: (1) a pivotal randomized cohort and (2) a valve-in-valve (ViV) cohort.

The objective of the pivotal randomized cohort is to evaluate the safety and effectiveness of the Navitor TAVI System for treating patients with symptomatic, severe native aortic stenosis who are considered intermediate or low risk for surgical mortality.

The Randomization Cohort will enroll approxmatly1500 subjects and will be randomized between the Navitor TAVI Implantation System (test arm) and any commercially available transcatheter aortic valve system (CAV) (control arm) in a 1:1 ratio.

The ViV cohort will be conducted as a separate prospective, multicenter, open label, two-group registry within the ENVISION IDE trial. A total of 250 subjects deemed to be at high or greater risk for open surgical therapy will be enrolled concurrently across two separate groups: 125 subjects undergoing transcatheter Aortic Valve-in-Surgical Aortic Valve replacement (TAV-in-SAV) and 125 subjects undergoing Transcatheter Aortic Valve-in-Transcatheter Aortic Valve replacement (TAV-in-TAV).

ELIGIBILITY:
Key Inclusion Criteria:

1. Subject who is deemed to be at intermediate or low risk for open surgical aortic valve replacement:

   1. Intermediate risk: estimated risk of overall surgical mortality ≥ 3% and < 8% at 30 days
   2. Low risk: estimated risk of overall surgical mortality < 3% at 30 days Estimated risk of overall surgical mortality includes consideration of the Society of Thoracic Surgeons (STS) risk score, overall clinical status, and other clinical co-morbidities unmeasured by the risk calculator
2. New York Heart Association (NYHA) Functional Classification of II, III, or IV
3. Degenerative aortic valve stenosis

Key Exclusion Criteria:

1. In the opinion of the Investigator, life expectancy is less than 2 years
2. Evidence of an acute myocardial infarction [defined as ST-segment elevation myocardial infarction (STEMI) or non-ST-segment elevation myocardial infarction (NSTEMI) with acute ischemia symptoms and troponin elevation] within 30 days prior to index procedure
3. Untreated clinically significant coronary artery disease requiring revascularization
4. Any percutaneous coronary or peripheral interventional procedure performed within 30 days prior (except pacemaker or implantable cardioverter defibrillator (ICD) implant) to index procedure or planned within 30 days following the index procedure
5. Blood dyscrasias as defined: leukopenia (WBC < 3000 mm3), acute anemia (Hb < 9 g/dL), thrombocytopenia (platelet count < 50,000 cells/mm³); history of bleeding diathesis or coagulopathy
6. Active peptic ulcer or upper GI bleeding within 3 months prior to index procedure that would preclude anticoagulation
7. Recent (within 6 months prior to index procedure date) cerebrovascular accident (CVA) or a transient ischemic attack (TIA)
8. Renal insufficiency (creatinine > 3.0 mg/dL or eGFR < 30 ml/min/1.73m2) and/or end stage renal disease requiring chronic dialysis
9. Hostile chest or conditions or complications from prior surgery that would make the subject be considered high surgical risk (i.e., mediastinitis, radiation damage, abnormal chest wall, porcelain aorta, adhesion of aorta or internal mammary artery to sternum, etc.)
10. Significant frailty as determined by the heart team (after objective assessment of frailty parameters) that would indicate high or extreme surgical risk
11. Mixed aortic valve disease (aortic stenosis and aortic regurgitation with predominant aortic regurgitation 3-4+)
12. Aortic valve is a unicuspid or bicuspid valve as verified by echocardiography or CT.
13. Severe ventricular dysfunction with LVEF < 30% as measured by resting echocardiogram
14. Pre-existing prosthetic heart valve or other implant (such as prosthetic ring or transcatheter edge-to-edge repair (TEER) clip) in any valve position
15. Severe circumferential mitral annular calcification (MAC) which is continuous with calcium in the left ventricular outflow tract (LVOT)
16. Severe (greater than or equal to 3+) mitral regurgitation or severe mitral stenosis
17. Minimum access vessel diameter of < 5.0 mm for small FlexNav Delivery System and < 5.5 mm for large FlexNav Delivery System
18. Eccentricity ratio of the annulus < 0.73

Additional Exclusion Criteria for Pivotal Randomized Cohort

1. Hostile Chest or conditions or complications from prior surgery that would make the subject be considered high surgical risk
2. Significant frailty as determined by the heart team (after objective assessment of frailty parameters) that would indicate high or extreme surgical risk
3. Mixed aortic valve disease
4. Aortic valve is a unicuspid or bicuspid valve as verified by echocardiography or CT
5. Inadequate aortic valve calcification
6. Pre-existing prosthetic heart valve or other implant (such as prosthetic ring or transcatheter edge-to-edge repair (TEER) clip) in any valve position

Additional Exclusion Criteria for ViV Cohort

1. Failing valve has moderate or greater paravalvular regurgitation.
2. Known severe prosthesis-patient mismatch
3. Failing valve is unstable, rocking, or not structurally intact.
4. Patient has a pre-existing prosthetic heart valve or other implant (such a prosthetic ring with a rigid support structure or transcatheter edge-to-edge repair clip) in any valve position other than aortic.
5. Bioprosthetic valve diameter that would not accommodate implantation of the Navitor Valve.
6. Increased risk of coronary obstruction by prosthetic leaflets of the index valve

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2036-04 (Estimated)

PRIMARY OUTCOMES:
Composite of all-cause mortality or all stroke | At 12 months post-procedure
  Number of patients that had any of the outcome events.

CONTACTS AND LOCATIONS:
Overall Officials: Barathi Sethuraman, Study Director — Abbott Structural Heart; Michael Reardon, MD, Study Chair — The Methodist Hospital Research Institute; Azeem Azeem, MD, Study Chair — Montefiore Medical Center; Bassem Chehab, MD, Principal Investigator — Ascension Via Christi Hospitals Wichita, Inc.; Ibrahim Sultan, MD, Principal Investigator — The University of Pittsburgh Medical Center
Locations (66):
- United States (60):
  - St. Joseph's Hospital & Medical Center, Phoenix, Arizona
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Kaiser Permanente Fontana Medical Center, Fontana, California
  - Southern California Permanente Medical Group - La Jolla, La Jolla, California
  - University of California at San Francisco, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Los Robles Regional Medical Center, Thousand Oaks, California
  - St. Joseph's Hospital & Medical Center, Denver, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - HCA Florida - JFK Hospital, Atlantis, Florida
  - HCA Florida Largo Hospital, Largo, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - HCA Florida Ocala Hospital, Ocala, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - The Queen's Medical Center, Honolulu, Hawaii
  - University of Chicago Medical Center, Chicago, Illinois
  - Endeavor Health, Evanston, Illinois
  - Northwestern Memorial Hospital, Evanston, Illinois
  - Ascension St. Vincent, Indianapolis, Indiana
  - Via Christi Regional Medical Center - St. Francis Campus, Wichita, Kansas
  - Ochsner Medical Center, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - MyMichigan Medical Center Midland, Midland, Michigan
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Morristown Medical Center, Morristown, New Jersey
  - Presbyterian Hospital, Albuquerque, New Mexico
  - Winthrop-University Hospital, Mineola, New York
  - New York University Langone Medical Center - Tisch Hospital, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Columbia University Medical Center/NYPH, New York, New York
  - Montefiore Medical Center - Moses Division, New York, New York
  - Mission Health & Hospitals, Asheville, North Carolina
  - East Carolina Heart Institute, Greenville, North Carolina
  - Christ Hospital, Cincinnati, Ohio
  - The Cleveland Clinic, Cleveland, Ohio
  - Ohio Health Research Institute, Columbus, Ohio
  - Hillcrest Medical Center, Tulsa, Oklahoma
  - Pinnacle Health System, Mechanicsburg, Pennsylvania
  - Allegheny General Hospital - ASRI, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Lankenau Institute for Medical Research, Wynnewood, Pennsylvania
  - North Central Heart, Sioux Falls, South Dakota
  - Baptist Memorial Hospital, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Ascension Texas Cardiovascular, Austin, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - Baylor Scott & White - The Heart Hospital Plano, Plano, Texas
  - Intermountain Health St George Regional Hospital, St. George, Utah
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Swedish Medical Center, Seattle, Washington
  - Aurora Medical Group, Milwaukee, Wisconsin
- Canada (6):
  - St. Paul's Hospital, Vancouver, British Columbia
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Institut de Cardiologie de Montreal (Montreal Heart Inst.), Montreal, Quebec
  - The Royal Victoria Hospital, Montreal, Quebec
  - Saint John Regional Hospital - New Brunswick Heart Centre, Saint John

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available to other researhers.